CLINICAL TRIAL: NCT06782997
Title: Performance of the Electroretinogram, Performed and Interpreted by an Advanced Practice Nurse, in the Screening for Diabetic Retinopathy.
Acronym: ERGDIAB
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PR25001
Record Dates: First submitted 2025-01-07; First posted 2025-01-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes mellitus; electroretinography; screening; diabetic retinopathy; advanced practice nurse
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — Electroretinography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetic Patients: Any diabetic hospital patient requiring screening for diabetic retinopathy
  Interventions: Device: Electroretinogram

INTERVENTIONS:
Device: Electroretinogram — Electroretinogram (RETevalTM devices, LKC Technologies) performed and interpreted by an advanced practice nurse compared to the gold standard (retinography) interpreted by an ophthalmologist

SUMMARY:
Diabetic retinopathy (DR) is a common microvascular complication of diabetes mellitus and the leading cause of preventable blindness in working-age individuals. Early screening for DR is a public health issue. The gold standard is fundoscopy interpreted by an ophthalmologist. In France, in 2020, it was estimated that one-third of diabetic patients had not seen an ophthalmologist in over two years. Recently, a portable electroretinogram (ERG), which provides a physiological and non-invasive assessment of retinal cell function, has been developed. It combines pupillary responses through an infrared-sensitive camera, the implicit time and the response amplitude to brief white light stimuli. The result is expressed as an overall score (DR score), considered abnormal if it is < 7 or > 23.4. The sensitivity of the ERG for screening diabetic retinopathy is estimated at 80%, and its specificity at 82%, compared to conventional imaging. Additionally, it has been shown that poor glycemic control is associated with an increase in implicit time in preclinical DR. This test could therefore detect earlier changes than imaging results. To date, it is not considered the gold standard in France. The investigators aim to test this hypothesis. The investigators propose a prospective, bi-center study to evaluate the performance of the ERG, performed and interpreted by an Advanced Practice Nurse (APN), compared to the gold standard of retinal imaging (retinography) interpreted remotely by an ophthalmologist.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a common microvascular complication of diabetes mellitus and the leading cause of preventable blindness in working-age individuals. Early screening for DR is a public health issue. The gold standard is fundoscopy interpreted by an ophthalmologist. In France, in 2020, it was estimated that one-third of diabetic patients had not seen an ophthalmologist in over two years. Recently, a portable electroretinogram (ERG), which provides a physiological and non-invasive assessment of retinal cell function, has been developed. It combines pupillary responses through an infrared-sensitive camera, the implicit time and the response amplitude to brief white light stimuli. The result is expressed as an overall score (DR score), considered abnormal if it is < 7 or > 23.4. The sensitivity of the ERG for screening diabetic retinopathy is estimated at 80%, and its specificity at 82%, compared to conventional imaging. Additionally, it has been shown that poor glycemic control is associated with an increase in implicit time in preclinical DR. This test could therefore detect earlier changes than imaging results. To date, it is not considered the gold standard in France. The investigators aim to test this hypothesis. The investigators propose a prospective, bi-center study to evaluate the performance of the ERG, performed and interpreted by an Advanced Practice Nurse (APN), compared to the gold standard of retinal imaging (retinography) interpreted remotely by an ophthalmologist.

The investigators' study will prospectively include adult patients with type 1 or type 2 diabetes mellitus and without know DR. These patients are followed in both study centers and both examinations (ERG and retinography) will be performed during the hospitalization for the evaluation of their diabetes and complications. Sensitivity and specificity of the ERG performed and interpreted by an APN will be compared to gold standard.

ELIGIBILITY:
Inclusion criteria:

* Patients > 18 years old
* With type 1 or type 2 diabetes mellitus
* No known diabetic retinopathy
* Affiliated to a social security system
* Attending the hospitals of Reims or Charleville Mézières in France during a hospitalization for the evaluation of their diabetes and complications

Exclusion criteria:

* Known diabetic retinopathy
* Ongoing pregnancy or within 3 months postpartum
* Recent cataract surgery (< 3 months)
* Photosensitive epilepsy
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 1 or type 2 diabetes mellitus and without know DR, followed in both study centers and hospitalized for the evaluation of their diabetes and complications.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the electroretinogram | during the patient's hospitalization, an average of 1 week
  Sensitivity of the electroretinogram, performed and interpreted by an advanced practice nurse, for screening diabetic retinopathy compared with the gold standard (retinography interpreted by an ophthalmologist).

SECONDARY OUTCOMES:
Specificity, positive predictive value and negative predictive value of the ERG | during the patient's hospitalization, an average of 1 week
  Specificity, positive predictive value and negative predictive value of the ERG performed and interpreted by an advanced practice nurse, for screening diabetic retinopathy compared with the gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France